CLINICAL TRIAL: NCT04999956
Title: Accuracy and Primary Stability in Immediate Implant Placement Using Dynamic Navigation or Freehand
Brief Title: Accuracy and Primary Stability in Immediate Implant Placement: Dynamic Navigation Versus Freehand
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH9H-2020-T122-2
Record Dates: First submitted 2021-07-29; First posted 2021-08-11 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Tooth Diseases
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic navigation (Experimental): Dental implant placement using a dynamic navigation system
  Interventions: Procedure: dynamic navigation surgery
- freehand (Sham Comparator): Dental implant placement using freehand technique
  Interventions: Procedure: freehand surgery

INTERVENTIONS:
Procedure: dynamic navigation surgery — immediate implant placement using dynamic navigation
  Arms: dynamic navigation
Procedure: freehand surgery — immediate implant placement using freehand surgery
  Arms: freehand

SUMMARY:
Prosthetic-driven immediate implant placement for optimal aesthetic restoration has been increasing in demand during the last decades but requires higher accuracy. Dynamic navigation has been reported better implant positioning. However, dynamic navigation's application to immediate implant placement has not been studied, and its exact role is still needed to be investigated further. Besides, implant insertion angle may influence primary stability, which is a prerequisite in achieving osseointegration, while dynamic navigation can precisely control angle and position. Therefore, the investigators designed a randomized controlled clinical trial study to verify the clinical efficacy of dynamic navigation and freehand in immediate implant placement. Patients will then be followed up one year after delivery of the crown to assess additional parameters.

DETAILED DESCRIPTION:
Prosthetic-driven immediate implant placement for optimal aesthetic restoration has been increasing in demand during the last decades but requires higher accuracy. Dynamic navigation has been reported better implant positioning. However, dynamic navigation's application to immediate implant placement has not been studied, and its exact role is still needed to be investigated further. Besides, implant insertion angle may influence primary stability, which is a prerequisite in achieving osseointegration, while dynamic navigation can precisely control angle and position. Therefore, the investigators designed a randomized controlled clinical trial study to verify the clinical efficacy of dynamic navigation and freehand in immediate implant placement. Patients will then be followed up one year after delivery of the crown to assess additional parameters.

These will include the assessment of soft tissue inflammation, cytokine concentrations, microbiome, stability of the buccal bone plate.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and in good health;
2. The maxillary incisor that cannot be retained due to non-periodontitis;
3. The buccal bone plate is complete;
4. No acute infection;
5. The extraction socket have at least 3-5 mm apical bone.

Exclusion Criteria:

1. General contraindications of oral implant surgery (such as immunodeficiency, long-term use of corticosteroids);
2. Treatments or diseases that may affect bone tissue metabolism (for example, taking bisphosphonates or receiving local radiotherapy);
3. Periodontitis history or uncontrolled periodontitis. Bleeding of probing (BOP) positive site ≥ 10%, or probing depth (PD) ≥ 4mm;
4. Heavy smokers or previous heavy smoking history (quit smoking time <5 years or> 20 cigarettes per day);
5. Refuse to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | before surgery to after surgery one week
  Taking cone-beam computed tomography (CBCT). The deviation between the planned implant and the actual implant were measured by Computer Assisted Dental Implant Precision System (Dcarer, Suzhou, China) as follows: (1) At least four feature points (like tooth cusps or bone pits) were selected in preoperative and postoperative CBCT for rough registration. (2) Feature surface circles in preoperative CBCT were selected, and then a mathematical algorithm displayed a similar feature surface circle in postoperative CBCT. The algorithm registered thousands of points in these two circles via conventional iso-surface thresholding technology. The software calculated registration error automatically. (3) Finally, the planned and actual implant were identified, and the deviation would be automatically calculated.
Peri-implant soft tissue health | 12-months follow-up after delivery of crown
  Assessment of tissue health according to the definition of the 2017 International Classification. Berglundh et al.

SECONDARY OUTCOMES:
Insetion torque value (ITV) | surgery day
  A general method to to detect primary stability roughly. The ITV were evaluated by a wrench (Straumann, Waldenburg, Switzerland) at the time of implant placement. The investigator record the number of scale. Being equal to or greater than 35N is a ideal primary stability.
Implant Stability Quotient (ISQ) | surgery day
  A device to detect primary stability precisely. A Smartpeg was screwed into each implant, and resonance frequency analysis (RFA) was performed using Osstell Mentor (Osstell/Integration Diagnostics, Goteborg, Sweden). ISQ were recorded in the buccal and the palatal directions three times and averaged. <60 represents low stability; 60-70 represents medium stability; higher than 70 represents high stability.
Esthetic appearance of the dental crown | 12-months follow-up after delivery of the crown
  PES-WES Score assessed using the Belser criteria
Patient satisfaction | 12-months follow-up after delivery of crown
  Assessed using a visual analogue scale (VAS=100mm, with 0=completely dissatisfied and 100 completely satisfied).
Peri-implant sulcus fluid Inflammation | 12-months follow-up after delivery of crown
  Cytokine concentrations determined by multiplex ELISA
Buccal bone changes | 12-months follow-up after delivery of crown
  Measurements performed on post-operative CBCT taken for routine follow-up
Implant microbiome | 12-months follow-up after delivery of crown
  16S microbiome analysis performed on submarginal biofilm taken with a sterile paper point

CONTACTS AND LOCATIONS:
Overall Officials: Junyu Shi, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (3):
- China (3):
  - Department of Oral and Maxillo-facial Implantology, Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Department of Oral and Maxillofacial Implantology, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided